CLINICAL TRIAL: NCT03213184
Title: Children's Respiratory and Environmental Workgroup (CREW)02
Brief Title: Children's Respiratory and Environmental Workgroup
Acronym: CREW02
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Chicago (Other); University of California, San Francisco (Other); Harvard School of Public Health (HSPH) (Other); University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0837; 1UG3OD023282 (NIH); A536700 (Other: UW Madison); SMPH\PEDIATRICS\PEDIATRICS (Other: UW Madison); Protocol V4.0, dated 11/13/18 (Other: HS-IRB, UW Madison); 5UH3OD023282-05 (NIH)
Record Dates: First submitted 2017-06-28; First posted 2017-07-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Asthma; Allergic Asthma; Allergies; Healthy
Keywords: Birth cohort; asthma; allergies
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples separated into plasma/serum aliquots and red blood cell/buffy coat
  * Urine
  * Stool
  * Nasal wash/blow/lavage
  * Nasal Brushing collected cells expanded in cell culture and cryopreserved
  * Baby teeth (dependent on number returned and amount of material needed for assay)
  * Hair and toenail clippings
  * Saliva
  * Home dust samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The environment during the prenatal period and in early life is a major contributor to the risk of developing childhood asthma. Birth cohort studies from single research centers have identified several factors that affect the risk for developing childhood asthma, including being exposed in early life to allergens, pollutants, viruses and bacteria, and psychosocial stress. Despite such advances, further progress in understanding the root causes of asthma have been hampered by the small size of previous studies, which makes it difficult to: 1) identify asthma risk factors with certainty, 2) know how environmental factors across the United States (U.S.) affect asthma, and 3) whether there are critical ages when pregnant mothers, infants and young children are particularly susceptible to these influences. Furthermore, different research groups tend to use different methods to study asthma, making it difficult to either compare or pool findings. One other challenge is that there are several types (i.e. phenotypes, endotypes) of childhood asthma, but these are poorly understood. To help overcome these challenges, investigators leading 12 asthma birth cohorts across the U.S. have established the Children's Respiratory Research Workgroup (CREW) consortium. CREW proposes to identify specific types of childhood asthma, develop an understanding of what early life environmental influences cause these different types of asthma and when, and identify targets for future efforts aimed at preventing childhood asthma.

DETAILED DESCRIPTION:
CREW is an NIH-funded project consisting of 12 individual U.S. birth cohorts and two scientific centers working together to identify phenotypes and causes of childhood asthma. CREW will include data from a large number of children (over 9,000 at birth, 6,000-7,000 who are still being followed, and at least 5,667 expected to enroll in CREW) and their families, with broad diversity in terms of ethnicity, family characteristics, neighborhoods and geographic locations. One of the primary goals of CREW is to put together sets of data and samples of participating cohorts to identify phenotypes of childhood asthma (i.e. specific subtypes of asthma that can be distinguished by clinical features such as natural history, triggers, exacerbation frequency, concurrent allergies, lung function, sex, etc). As we obtain mechanistic insights about personal and early life risk factors, we will connect asthma phenotypes with underlying causes and pathogenic mechanisms to define endotypes of childhood asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent guardian must be able to understand and provide informed consent or assent (if required).
2. Participation in one of the 10 cohorts that make up CREW.

Exclusion Criteria:

1. Inability or unwillingness of a participant to give informed consent or assent (if required) or comply with study protocol.
2. Past or current medical problems or findings from physical examination or laboratory testing which, in the opinion of the investigator or designee, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CREW consortium represent a diverse national sample of children and families recruited over the past 30 years into 12 early life and birth cohort studies that focused on asthma. The total combined study population is 8,985 at the time of birth. The study population is quite diverse in terms of current age (ages <1 through 36 years), date of recruitment (1980-2017), race/ethnicity, and risk of asthma. There is considerable variation in the geographic locations of participants, with representation from East Coast (Baltimore, Boston, New York City), Midwest (Cincinnati, Detroit, Madison, Marshfield), South (Nashville, St. Louis) and West (Tucson). Most children are healthy (control population) while some have asthma or some form of allergic disease.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in the first second (FEV1) | 7 years
  Spirometry, also known as FEV1, will be measured at all ages to asses level of asthma.

SECONDARY OUTCOMES:
Asthma Control Test (ACT) | 7 years
  Asthma symptoms of children leading to differing asthma severity (none, mild, moderate, severe) will be measured using the ACT questionnaire at all ages.
Immunoglobulin E (IgE) | 7 years
  Total IgE will be measured serologically and will be used to determine level of allergy in all ages over 7 years.

CONTACTS AND LOCATIONS:
Overall Officials: James Gern, MD, Principal Investigator — UW Madison; Daniel Jackson, MD, Principal Investigator — UW Madison
Locations (10):
- United States (10):
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UW Madison, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No